CLINICAL TRIAL: NCT00670865
Title: Automated Versus Conventional Hospital Discharge Summaries and Prescriptions: A Randomized Controlled Trial
Brief Title: Automated Versus Conventional Hospital Discharge Summaries and Prescriptions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: David Maslove, MD. Chief Medical Resident, St. Michael's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 07-364
Record Dates: First submitted 2008-04-07; First posted 2008-05-02 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2010-04

CONDITIONS: Patient Discharge; Continuity of Patient Care; Medical Records Systems, Computerized; Hospital Information Systems
Keywords: Hospitalization; Continuity of care; Discharge summary; Quality improvement; Medical records systems; Hospital information systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- eDischarge (Experimental): The eDischarge arm will consist of two teams on the General Internal Medicine ward at St. Michael's Hospital who have been randomly assigned to use the electronic discharge summary program.
  Interventions: Other: Electronic discharge summary system
- Traditional (No Intervention): The traditional arm will consist of two teams on the General Internal Medicine ward at St. Michael's Hospital who have been randomly assigned to use "traditional," dictated discharge summaries.

INTERVENTIONS:
Other: Electronic discharge summary system — The customized electronic discharge summary program will be used to generate patient discharge summaries.
  Arms: eDischarge

SUMMARY:
The purpose of this study is to determine whether a semi-automated electronic patient discharge summary program leads to increased community physician and housestaff satisfaction and patient outcomes as compared to conventional discharge reports.

DETAILED DESCRIPTION:
For patients hospitalized with an acute illness, the days following discharge constitute a critical period. Patients must adjust to changes in their medications, follow up with family doctors and other specialists and know what symptoms should prompt a return to hospital. The community physicians who follow them rely on information from their hospitalization to facilitate this transition, and provide continuity of care.

Communication between hospital and community physicians is essential to this process, and has traditionally been accomplished by a dictated discharge summary. Previous studies have shown that while dictated discharge summaries can be inaccurate, incomplete, or untimely, computer generated summaries are produced more quickly and accurately. Moreover, database-generated discharge summaries are preferred by physicians in the community.

We have designed a web-based computer program with quality assurance features that automatically generates timely discharge summaries. We aim to study this program over a 2 month period on our general medicine unit by means of a randomized controlled trial. Our hypothesis is that community physicians will prefer the computer generated summaries, over the standard dictated summaries. If effective, our system could be implemented more widely, and would stand to improve communication with community physicians, continuity of care, and patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization on General Internal Medicine ward at St. Michael's Hospital

Exclusion Criteria:

* Transfer to another service
* Death during admission
* Remains in hospital past dates specified in study protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2008-05; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Primary care physician satisfaction from satisfaction score assessment form with 100-mm visual analogue scale | Satisfaction score assessment form to be sent one week after patient's discharge from hospital. If form is not returned in 14 days, a reminder and second form will be sent.

SECONDARY OUTCOMES:
St. Michael's Hospital housestaff satisfaction from satisfaction score assessment form with 100-mm visual analogue scale | Housestaff will fill out form upon completion of the rotation during which the study has been performed
Completion of specialist outpatient workups at St. Michael's Hospital recommended during course of hospitalization | Within the first 30 days of patient's discharge from hospital
Patient visits to Emergency Room at St. Michael's Hospital | Within the first 30 days after patient's discharge from hospital
Patient/proxy care transition assessment through the use of the CTM-3. | Phone call made to patient or proxy one week after discharge. If patient/proxy is not reached, follow up calls will be made daily until patient/proxy is reached.
Prescribing errors as assessed by comparing discharge summary to inpatient record | Upon discharge
Patient readmissions to St. Michael's Hospital | Within 30 days of discharge

CONTACTS AND LOCATIONS:
Overall Officials: David M Maslove, MD, Principal Investigator — Unity Health Toronto; Chaim M Bell, MD, PhD, FRCPC, Principal Investigator — St. Michael's Hospital; University of Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] van Walraven C, Laupacis A, Seth R, Wells G. Dictated versus database-generated discharge summaries: a randomized clinical trial. CMAJ. 1999 Feb 9;160(3):319-26. PMID 10065073
- [Background] van Walraven C, Seth R, Austin PC, Laupacis A. Effect of discharge summary availability during post-discharge visits on hospital readmission. J Gen Intern Med. 2002 Mar;17(3):186-92. doi: 10.1046/j.1525-1497.2002.10741.x. PMID 11929504
- [Background] Kripalani S, LeFevre F, Phillips CO, Williams MV, Basaviah P, Baker DW. Deficits in communication and information transfer between hospital-based and primary care physicians: implications for patient safety and continuity of care. JAMA. 2007 Feb 28;297(8):831-41. doi: 10.1001/jama.297.8.831. PMID 17327525
- [Result] Maslove DM, Leiter RE, Griesman J, Arnott C, Mourad O, Chow CM, Bell CM. Electronic versus dictated hospital discharge summaries: a randomized controlled trial. J Gen Intern Med. 2009 Sep;24(9):995-1001. doi: 10.1007/s11606-009-1053-2. Epub 2009 Jul 16. PMID 19609623